CLINICAL TRIAL: NCT07159464
Title: Post Study Access of CSL312 (Garadacimab) for the Routine Prevention of Hereditary Angioedema (HAE) Attacks in Pediatric Participants (2-11 Years Old) With HAE Who Have Completed the CSL312_3003 Study
Brief Title: Post Study Access of CSL312 (Garadacimab) for Pediatric Participants With Hereditary Angioedema Who Have Completed the CSL312_3003 Study
Status: Available | Type: Expanded Access
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Other Study IDs: CSL312_5001
Record Dates: First submitted 2025-08-28; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Hereditary Angioedema (HAE)
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: CSL312 — Fully human immunoglobulin G subclass 4/lambda recombinant inhibitor monoclonal antibody administered subcutaneously (SC)
  Other Names: Garadacimab

SUMMARY:
This protocol for post study access allows pediatric participants (2-11 years old at the time of consent) with HAE who have completed study CSL312_3003 (NCT05819775) to continue treatment with CSL312 for routine prevention of HAE attacks. The continuing treatment with the study product will be administered under a Post Study Access program in accordance with the applicable laws and regulations, to be dictated by CSL Behring (Sponsor) and approved by the appropriate local/central Ethics Committees and all other competent authorities required by law, as applicable.

ELIGIBILITY:
Inclusion Criteria:

* Completion of treatment period in study CSL312_3003 (NCT05819775)
* The participant responded to CSL312 treatment with no or very limited number of HAE attacks during the CSL312_3003 study
* The participant experienced no clinically significant adverse effects associated with CSL312 treatment
* In the opinion of the treating physician, the participant continues to receive benefit from CSL312
* There is no other suitable alternative prophylactic treatment available at the time of consenting into the Post Study Access program

Exclusion Criteria:

* In the opinion of the treating physician, participant may not be compliant with the Protocol requirements
* Participant is 12 years or older at the time of consent
* In the opinion of the treating physician, other study medication of prophylaxis treatment of HAE may benefit the participant more than continuing treatment with CSL312
* Participant who is pregnant, breastfeeding, or not willing to cease breastfeeding

Max Age: 11 Years | Sex: All
Age Groups: Child